CLINICAL TRIAL: NCT03672734
Title: Observed Volume and pH of Gastric Contents in Patients Undergoing Gynecologic Laparoscopic Surgery During Emergence From General Anesthesia
Brief Title: Volume and pH of Gastric Contents in Patients Undergoing Gynecologic Laparoscopic Surgery During Emergence From General Anesthesia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Warunee Boayam, Department of Anesthesiology, Faculty of Medicine Siriraj Hospital, Mahidol university, Siriraj Hospital
Other Study IDs: 328/2561(EC3)
Record Dates: First submitted 2018-08-31; First posted 2018-09-14 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2018-09

CONDITIONS: General Anesthesia
Keywords: pH gastric contents; laparoscopic surgery; pH stomach; volume gastric content

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Complications during general anesthesia,induction period: difficult airway, hypotension, upper airway obstruction, laryngospasm, pulmonary aspiration Maintenance period: hypotension, hypertension, awareness, bronchospasm, pulmonary aspiration.

Emergence period: delayed emergence, upper airway obstruction, pulmonary aspiration.

Pulmonary aspiration occur all ranges of general anesthesia. Because the patients can not protected themselves due to anesthetic medication, example: volatile agent, opioid.This can cause decrease consciousness, delayed gastric emptying time. Incidence of pulmonary aspiration was 1 : 900 - 1 : 10,000 of general of anesthesia (induction 20%, emergence 80%), Anesthesia Service in Siriraj Hospital (2017) 6: 25,000 case Pathophysiology of pulmonary aspiration.

Pulmonary aspiration is defined as inhalation of oropharynx or stomach contents through the larynx to low respiratory tract. Aspiration pneumonitis is the inflammation of the lung caused by aspirating or inhaling irritants (Mendelson's syndrome).

Gastric acid is a digestive fluid formed in the stomach and is composed of hydrochloric acid, potassium chloride, and sodium chloride.The highest concentration of gastric acid is 140-160 mEq/L. The pH of gastric acid is 1.5-3.5 in the human stomach lumen.

Risk factors for increased gastric contents: full stomach, delayed gastric emptying, incompetent lower esophageal sphincter, lithotomy position, laparoscopy, length of surgery more than 2 hr., difficult airway.

This study observed Volume and pH of Gastric Contents in Patients undergoing Gynecologic Laparoscopic Surgery during Emergence from General Anesthesia.

DETAILED DESCRIPTION:
The study was approved from the Siriraj Institutional Review Board (Si-IRB), COA (Certificate of Analysis):Si437/2018 and was written informed consent was obtained from all subjects. The study was conducted at the Department of Siriraj Obstetrics and Gynecology.

A total of 100 patients were enrolled in the study between September 2018 and 2019. All patients underwent general anesthesia for elective gynecologic laparoscopic surgery. Inclusion criteria were elective Cases, laparoscopic surgery, age 18-65 year,BMI<30kg/sq.m. Exclusion criteria were emergency Case, full stomach. Withdrawal or termination criterion was the difficult inserted orogastric tube.

On the day of surgery, participants signed the informed consent. Record data consisted of NPO time, premedication drug, BMI, having intravenous fluid. All patients underwent general anesthesia after application of standard monitors, anesthesia was induced with fentanyl 1-2 mcg/kg. or morphine 0.1-0.2 mg/kg., propofol 1.5-2.5 mg/kg.,nimbex 1-1.5 mg/kg or atracurium 0.6 mg/kg. Anesthesia was maintained with sevoflurane, air, o2.

Gastric volume and PH were measured with PH meter, measured at 1hr. intervals until the end of surgery. Intraoperative, record medication for reduced gastric volume or PH.

Postoperative, data were record nausea or vomiting, medication requirements.

ELIGIBILITY:
Inclusion Criteria:

* ASA class 1-2,
* 18-65 years old,
* Laparoscopic surgery,
* BMI<30kg/sq.m.

Exclusion Criteria:

* Difficult inserted orogastric tube.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients underwent gynecologic laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-09-20 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
pH of Gastric Contents | 6 hours
  After general anesthesia, the investigator will insert an orogastric tube to drain the all the gastric secretion until the end of surgery. The pH of the content will be measured at the end of the operation.

SECONDARY OUTCOMES:
Volume of Gastric Content | 6 hours
  After general anesthesia, the investigator will insert an orogastric tube to drain the all the gastric secretion until the end of surgery. The volume of the content (mL.) will be measured at the end of the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Warunede Buayam, B.NS, Study Director — Department of Anesthesiology, Faculty of Medicine, Siriraj hospital
Locations (1):
- Waerunee Boayam, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perlas A, Chan VW, Lupu CM, Mitsakakis N, Hanbidge A. Ultrasound assessment of gastric content and volume. Anesthesiology. 2009 Jul;111(1):82-9. doi: 10.1097/ALN.0b013e3181a97250. PMID 19512861
- [Background] Ouanes JP, Bicket MC, Togioka B, Tomas VG, Wu CL, Murphy JD. The role of perioperative chewing gum on gastric fluid volume and gastric pH: a meta-analysis. J Clin Anesth. 2015 Mar;27(2):146-52. doi: 10.1016/j.jclinane.2014.07.005. Epub 2014 Nov 28. PMID 25442242
- [Background] Schmidt AR, Buehler P, Seglias L, Stark T, Brotschi B, Renner T, Sabandal C, Klaghofer R, Weiss M, Schmitz A. Gastric pH and residual volume after 1 and 2 h fasting time for clear fluids in childrendagger. Br J Anaesth. 2015 Mar;114(3):477-82. doi: 10.1093/bja/aeu399. Epub 2014 Dec 13. PMID 25501720
- [Background] Phillips S, Liang SS, Formaz-Preston A, Stewart PA. High-risk residual gastric content in fasted patients undergoing gastrointestinal endoscopy: a prospective cohort study of prevalence and predictors. Anaesth Intensive Care. 2015 Nov;43(6):728-33. doi: 10.1177/0310057X1504300610. PMID 26603797
- [Background] Splinter WM. From the Journal archives: gastric fluid volume and pH in elective patients following unrestricted oral fluid until three hours before surgery. Can J Anaesth. 2014 Dec;61(12):1126-9. doi: 10.1007/s12630-014-0220-z. Epub 2014 Aug 15. No abstract available. PMID 25125250
- [Background] Goudra BG, Singh PM, Carlin A, Manjunath AK, Reihmer J, Gouda GB, Ginsberg GG. Effect of Gum Chewing on the Volume and pH of Gastric Contents: A Prospective Randomized Study. Dig Dis Sci. 2015 Apr;60(4):979-83. doi: 10.1007/s10620-014-3404-z. Epub 2014 Nov 2. PMID 25362513
- [Background] Ong BY, Palahniuk RJ, Cumming M. Gastric volume and pH in out-patients. Can Anaesth Soc J. 1978 Jan;25(1):36-9. doi: 10.1007/BF03006781. PMID 23891
- [Background] Gouda BB, Lydon AM, Badhe A, Shorten GD. A comparison of the effects of ranitidine and omeprazole on volume and pH of gastric contents in elective surgical patients. Eur J Anaesthesiol. 2004 Apr;21(4):260-4. doi: 10.1017/s0265021504004028. PMID 15109187
- [Background] Gombar S, Kiran S, Gupta M, Gombar K, Chhabra B. Preanaesthetic oral ranitidine, omeprazole and metoclopramide for modifying gastric fluid volume and pH. Can J Anaesth. 1994 Sep;41(9):879-80. doi: 10.1007/BF03011614. No abstract available. PMID 7955016
- [Background] Boulay K, Blanloeil Y, Bourveau M, Geay G, Malinovsky JM. Effects of oral ranitidine, famotidine and omeprazole on gastric volume and pH at induction and recovery from general anaesthesia. Br J Anaesth. 1994 Oct;73(4):475-8. doi: 10.1093/bja/73.4.475. PMID 7999487
- [Background] Chang KK, Jawan B, Fung ST, Lee JH. Effect of preoperative fasting time on gastric volume and pH. Ma Zui Xue Za Zhi. 1989 Jun;27(2):149-52. PMID 2796624
- [Background] Haavik PE, Soreide E, Hofstad B, Steen PA. Does preoperative anxiety influence gastric fluid volume and acidity? Anesth Analg. 1992 Jul;75(1):91-4. doi: 10.1213/00000539-199207000-00017. PMID 1535490
- [Background] Maltby JR, Lewis P, Martin A, Sutheriand LR. Gastric fluid volume and pH in elective patients following unrestricted oral fluid until three hours before surgery. Can J Anaesth. 1991 May;38(4 Pt 1):425-9. doi: 10.1007/BF03007577. PMID 2065409
- [Background] Noakes TD, Rehrer NJ, Maughan RJ. The importance of volume in regulating gastric emptying. Med Sci Sports Exerc. 1991 Mar;23(3):307-13. PMID 1875801
- [Background] Goetze O, Treier R, Fox M, Steingoetter A, Fried M, Boesiger P, Schwizer W. The effect of gastric secretion on gastric physiology and emptying in the fasted and fed state assessed by magnetic resonance imaging. Neurogastroenterol Motil. 2009 Jul;21(7):725-e42. doi: 10.1111/j.1365-2982.2009.01293.x. Epub 2009 Apr 1. PMID 19344341
- [Background] Brocks K, Jensen JS, Schmidt JF, Jorgensen BC. Gastric contents and pH after oral premedication. Acta Anaesthesiol Scand. 1987 Jul;31(5):448-9. doi: 10.1111/j.1399-6576.1987.tb02600.x. PMID 3630589